CLINICAL TRIAL: NCT02596399
Title: A PHASE I, RANDOMIZED, DOUBLE-BLIND,PLACEBO-CONTROLLED, SINGLE-ASCENDING DOSE STUDY TO INVESTIGATE THE SAFETY,TOLERABILITY, AND PHARMACOKINETICS OF DSTA4637S IN HEALTHY VOLUNTEERS
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of DSTA4637S in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV29259
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteers; DSTA4637S

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- DSTA4637S (Experimental)
  Interventions: Drug: DSTA4637S
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DSTA4637S — Participants will receive DSTA4637S intravenously on Day 1.
  Arms: DSTA4637S
Drug: Placebo — Participants will receive placebo matched to DSTA4637S intravenously on Day 1.
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-ascending dose study in healthy volunteers, enrolled at a single site in the United States to investigate the safety, tolerability, and pharmacokinetics of DSTA4637S.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Able to comply with the study protocol, in the investigator's judgment
* Body mass index (BMI) between 18 and 32 kilogram per square meters (kg/m^2), inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs
* Clinical laboratory evaluations should be within the reference range for the test laboratory unless deemed not clinically significant by the investigator and Sponsor
* Willing to abstain from the use of drugs of abuse through completion of the study
* Willing to abstain from use of over the counter, herbal or prescription medications/products from 14 days prior to Day 1 through completion of the study, unless deemed acceptable by the investigator and Sponsor
* Agreeable to, and deemed able to (by the investigator), comply with requirements of the study, including the follow-up period
* Willing to abstain from consumption of alcohol-based products from 72 hours prior to Day 1 until Phase 1 unit check-out on Day 3 and for 72 hours prior to each follow-up visit
* For women of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use non-hormonal contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 85 days after the last dose of study drug
* For men, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined in the study protocol

Exclusion Criteria:

* Any diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that in the opinion of the investigator or Sponsor contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications
* Use of tobacco, electronic cigarettes, personal vaporizer or electronic nicotine delivery systems (positive history within 3 months before initiation of dosing on Day 1)
* Received any vaccine within 14 days prior to screening
* Pregnant or lactating, or intending to become pregnant within 3 months after screening
* Positive serum pregnancy test result at screening or Day −1
* Received oral antibiotics within 4 weeks before initiation of dosing on Day 1, or intravenous antibiotics within 8 weeks before initiation of dosing
* Hospitalization within 4 weeks before initiation of dosing
* Positive for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody
* History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine, and crack) within 1 year prior to screening
* Positive drug screen at screening or Day -1
* History of anaphylactic or hypersensitivity drug reaction, unless approved by the investigator and Sponsor
* Blood transfusion within 8 weeks prior to screening
* History of malignancy within 10 years of screening except completely excised basal cell carcinoma or squamous cell carcinoma of the skin
* Donation of plasma (greater than or equal to [>=] 500 milliliter [mL]) within 7 days prior to study drug administration
* Donation or loss of whole blood (excluding the volume of blood that will be drawn during screening procedures) as follows: 50-499 mL of whole blood within 30 days or greater than (>) 499 mL of whole blood within 56 days prior to study drug administration
* Hemoglobin <128 gram per liter (g/L) (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females) at screening
* Poor peripheral venous access
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, evidence of prior myocardial infarction
* Exposure to any biological therapy or investigational biological agent within 90 days prior to the screening evaluation or have received any other investigational treatment 30 days prior to the screening evaluation (or within 5 half-lives of the investigational product, whichever is greater)
* Any history of hypersensitivity or allergy to rifampin or other rifamycin analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-29 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with at least 1 Adverse Event (AE) | Up to Day 85

SECONDARY OUTCOMES:
Concentration of analytes of DSTA4637S in plasma and serum | Up to Day 85
Concentration of anti-therapeutic antibodies (ATA) to DSTA4637S | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA International Clinical Pharmacology Center (EDS US Clinic), Lenexa, Kansas, United States

REFERENCES:
- [Derived] Peck M, Rothenberg ME, Deng R, Lewin-Koh N, She G, Kamath AV, Carrasco-Triguero M, Saad O, Castro A, Teufel L, Dickerson DS, Leonardelli M, Tavel JA. A Phase 1, Randomized, Single-Ascending-Dose Study To Investigate the Safety, Tolerability, and Pharmacokinetics of DSTA4637S, an Anti-Staphylococcus aureus Thiomab Antibody-Antibiotic Conjugate, in Healthy Volunteers. Antimicrob Agents Chemother. 2019 May 24;63(6):e02588-18. doi: 10.1128/AAC.02588-18. Print 2019 Jun. PMID 30910894